CLINICAL TRIAL: NCT06800716
Title: A Prospective Study of Recovery Mechanisms in Heart Transplant Eligible Patients With Cardiogenic Shock on Impella 5.5 Support
Brief Title: Impella Reverse Remodeling in End-Stage Heart Failure
Status: Recruiting | Type: Observational
Sponsor: Columbia University (Other)
Collaborators: Abiomed Inc. (Industry)
Responsible Party: Principal Investigator, Adil A Yunis, MD, Assistant Professor of Medicine, Columbia University
Other Study IDs: AAAV1201
Record Dates: First submitted 2025-01-08; First posted 2025-01-30 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Heart Failure; Cardiomyopathy
Keywords: cardiogenic shock and transplant; impella; LVAD
MeSH Terms: conditions — Heart Failure; Cardiomyopathies; Shock, Cardiogenic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Cardiac myocardium samples from the explanted heart of the transplant recipient.
  Serum samples from the transplant recipient.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (1):
- Decompensated patients on the waitlist for heart transplantation: Study participants will receive Impella 5.5 LVAD for treatment of cardiogenic shock and transplant listing as standard of care. Clinical data and serum laboratory including blood counts, end-organ function, nutritional parameters will be collected prospectively from medical records. Participants are required to complete an assessment a 6-minute walk, and hand grip strength test.

SUMMARY:
This observational study is being done to learn more about heart attack recovery in patients supported with the Impella 5.5 left ventricular assist device (LVAD) as part of their standard of care. There are three stages in this study: screening, treatment and post treatment. There will be two phases of enrollment: First phase will enroll 10 patients; second phase will enroll an additional 40 patients. Approximately 50 participants will take part in the study at Columbia University Irving Medical Center.

Participation in this research is expected to last approximately 14 months. This time estimate includes a screening period for about 1- 3 days, treatment period of 40 days and post treatment follow-up period for 1 year. Data will be collected through 1- year after heart transplant. Clinical data (medical history, vital signs, laboratory assessments) from medical records, to perform functional testing, and to obtain blood and discarded heart tissue fromfor the purpose of this research study.

Participants will be asked to share their records for echocardiography, right heart catheterization, laboratory data and clinical information. Participants are required to complete an assessment a 6-minute walk, and hand grip strength test.

DETAILED DESCRIPTION:
Percutaneous endovascular mechanical circulatory support (MCS) devices have been increasingly utilized in patients on the waitlist for heart transplantation in the new heart allocation system. However, the number of patients recovering from heart failure and delisted from cardiac transplantation has declined in the new heart allocation system. While significant research has been performed on myocardial recovery with durable left ventricular assist device (LVAD) support, natural course and mechanistic basis of reverse remodeling on percutaneous endovascular MCS remains unknown. The primary objective of this prospective, observational, single-center study is to evaluate whether mechanical circulatory support with Impella 5.5 LVAD in decompensated patients on the waitlist for heart transplantation results in left ventricular reverse remodeling and improvement in end-organ function within 14 days of initiating support. Phenotypic data including clinical information, echocardiography, and hemodynamics will be serially obtained in participants before and after Impella 5.5 LVAD placement. Paired serum samples (pre- and post- Impella support) will be obtained for proteomic analysis. Cardiac tissue samples will be collected at the time of cardiac transplantation for histopathological analysis as well as RNA-sequencing. Candidate genes and proteins of reverse remodeling will be validated using quantitative polymerase chain reaction (qPCR) and Western Blotting. This study will definitively establish the natural course of reverse remodeling in patients with chronically failing ventricles on Impella 5.5 support and determine molecular signals and novel biomarkers of myocardial recovery in this growing population. Data obtained from this study will help determine which patients should pursue recovery pathway as opposed to transplant.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Dilated cardiomyopathy (LVEDD > 5.5 cm and LVEF <25%)
* Indication for temporary mechanical circulatory support therapy with Impella 5.5 LVAD as a bridge to transplant or bridge to transplant decision based on treating physician's discretion

Exclusion Criteria:

* Intra-aortic balloon pump (IABP) use for more than 7 days at the time of Impella 5.5 implantation
* Percutaneous mechanical circulatory support device, extracorporeal membrane oxygenation (ECMO) or paracorporeal ventricular assist device (VAD) support prior to Impella 5.5 implantation
* Congenital heart disease
* Restrictive or hypertrophic Cardiomyopathy including hypertrophic obstructive cardiomyopathy (HOCM) Amyloidosis, and Sarcoidosis
* Evidence of acute myocarditis by endomyocardial biopsy
* Prior heart transplantation
* Mechanical aortic / mitral valve
* Patient with known aortic diseases such as Marfan-Syndrome, Morbus Erdheim-Gsell or others
* Left Ventricular thrombus
* Left Ventricular rupture
* Cardiac tamponade
* Presence of an Atrial or Ventricular Septal Defect
* Severe right ventricular (RV) Failure requiring mechanical RV support
* Severe peripheral vascular disease precluding placement of the Impella System
* Recent stroke resulting in significant neurological deficit
* Hypercoagulable disease precluding device implantation
* Severe thrombocytopenia (<50,000)
* Contraindication to anticoagulation
* Suspected or known pregnancy or lactating women
* Subject belongs to a vulnerable population

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Inpatients at Columbia University Irving Medical Center, who are waitlisted for heart transplant with a clinical indication for Impella 5.5 left ventricular assist device (LVAD) placement.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-12-04 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
Change in Left Ventricular Ejection Fraction (LVEF) | Baseline and approximately Day 40
  A change in echocardiographic index will be evaluated by measuring a change in LVEF before and after Impella support at minimal pump setting.
Change in Left Ventricular End-Diastolic Diameter (LVEDD) | Baseline and approximately Day 40
  A change in echocardiographic index will be evaluated by measuring a change in LVEDD before and after Impella support at minimal pump setting.
Change in Cardiac Index | Baseline and approximately Day 40
  A change in hemodynamics will be evaluated by measuring a change in cardiac index before and after Impella support at minimal pump speed setting (P2).
Change in Pulmonary Capillary Wedge Pressure | Baseline and approximately Day 40
  A change in hemodynamics will be evaluated by measuring a change in Pulmonary Capillary Wedge Pressure before and after Impella support at minimal pump speed setting (P2).

SECONDARY OUTCOMES:
Transplant Waitlist Outcome | 14 months
  The transplant waitlist outcome will be evaluated and the number of participants who die, are delisted due to worsening clinical condition, are transplanted, or are delisted for recovery will be reported.
Number of Participants Escalated | 14 months
  Number of participants escalated to extracorporeal membrane oxygenation (ECMO) or other temporary/durable mechanical circulatory support (MCS).
Waitlist time on Impella Support | 14 months
  Waitlist time on Impella support measured in days from the date of Impella insertion to heart transplantation or other waitlist end-point.
Change in aminoterminal pro B-type natriuretic peptide (NT-proBNP) | Baseline and approximately Day 40
  Change in NT-proBNP levels collected from blood samples and measured in pg/mL.
Change in Blood Urea Nitrogen (BUN) | Baseline and approximately Day 40
  Change in BUN levels collected from blood samples and measured in mg/dL.
Change in Estimated Glomerular Filtration Rate (eGFR) | Baseline and approximately Day 40
  Change in eGFR collected from blood samples and measured in mL/min/1.73m^2.
Change in Cystatin C | Baseline and approximately Day 40
  Change in Cystatin C collected from blood samples and measured in mg/L.
Change in Total Bilirubin | Baseline and approximately Day 40
  Change in Total Bilirubin collected from blood samples and measured in mg/dL.
Change in Aspartate Aminotransferase (AST) | Baseline and approximately Day 40
  Change in AST collected from blood samples and measured in U/L.
Change in Alanine Aminotransferase (ALT) | Baseline and approximately Day 40
  Change in ALT collected from blood samples and measured in U/L.
Change in International Normalized Ratio (INR) | Baseline and approximately Day 40
  Change in INR collected from blood samples. INR is a ratio and has no units of measure.
Change in Hemoglobin | Baseline and approximately Day 40
  Change in hemoglobin levels collected from blood samples and measured in g/L.
Change in Platelet Count | Baseline and approximately Day 40
  Change in platelet count collected from blood samples and measured in pl/μL.
Change in Lactate dehydrogenase (LDH) | Baseline and approximately Day 40
  Change in LDH collected from blood samples and measured in U/L.
Change in Plasma Free Hemoglobin | Baseline and approximately Day 40
  Change in plasma free hemoglobin collected from blood samples and measured in mg/dL.
Change in Prealbumin | Baseline and approximately Day 40
  Change in prealbumin collected from blood samples and measured in mg/dL.
Change in Albumin | Baseline and approximately Day 40
  Change in albumin collected from blood samples and measured in mg/dL.
Change in C-Reactive Protein (CRP) | Baseline and approximately Day 40
  Change in CRP collected from blood samples and measured in mg/L.
Change in Erythrocyte Sedimentation Rate (ESR) | Baseline and approximately Day 40
  Change in ESR collected from blood samples and measured in mm/hr.
Change in Procalcitonin | Baseline and approximately Day 40
  Change in procalcitonin collected from blood samples and measured in ng/mL.
Change in HLA Allosensitization Profile | Baseline and approximately Day 40
  Change in the HLA allosensitization profile. Allosensitization is the presence of circulating antibodies against human leukocyte antigens and nonhuman leukocyte antigens.
Change in Vasoactive-Inotropic Score (VIS) | Baseline and approximately Day 40
  Vasoactive-Inotropic Score (VIS) is calculated with the following formula: VIS = dopamine (µg/kg/min) + dobutamine (µg/kg/min) + 100 × epinephrine (µg/kg/min) + 100 × norepinephrine (µg/kg/min) + 10 × milrinone (µg/kg/min) + 10,000 × vasopressin (units/kg/min). Scores range from 0 to no upper limit, with a higher score indicating a worse outcome.
Six Minute Walk Test (6MWT) | 14 months
  The 6MWT is a measure of performance that assesses the distance walked in six minutes measured in meters. the 6MWT will be conducted in the Cardiac Care Unit (CCU) on device support.
Change in Upper Extremity Hand Strength | 14 months
  Change in upper extremity strength measured by Handgrip dynamometry in kilograms.
Units of Blood Used During Heart Transplant | Day of Transplant (Approximately Day 40)
  Units of red blood cells, cryoprecipitate, fresh frozen plasma, and platelets used during transplant.
Primary Graft Failure | 14 months
  The number of participants with primary graft failure after heart transplantation. Graft failure defined as left ventricular ejection fraction of <40%.
Early Transplant Rejection | 14 months
  The number of participants with early transplant rejection. Early transplant rejected defined as an episode of rejection within the first 3 months of transplant.
AlloMap Score | After Transplant, approximately Day 40
  AlloMap score after heart transplantation. AlloMap measures the risk of acute cellular rejection. Scores range from 0 - 40 with higher score indicating a worse outcome.
Allosure Score | After Transplant, approximately Day 40
  Allosure score after heart transplantation. Allosure measures the risk of rejection in heart transplant recipients. Scores range from a lower limit of < 0.04 and above with a higher score indicating a worse outcome.
Post-Transplant Length of Stay | Up to 14 months (approximately 420 days)
  Post-transplant length of hospital stay measured in days and assessed for up to 14 months.

CONTACTS AND LOCATIONS:
Overall Officials: Adil Yunis, MS, Principal Investigator — Columbia University
Locations (1):
- Columbia University, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided